CLINICAL TRIAL: NCT04550702
Title: Predictor for Re-treatment of Overactive Bladder Syndrome After Discontinuation of Mirabegron Treatment for Female Overactive Bladder Syndrome
Brief Title: Predictors for Retreatement of OAB After DC Mirabegron
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202006091RIND
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-07

CONDITIONS: Recurrence of Overactive Bladder Syndrome
Keywords: overactive bladder syndrome; beta-3 agonist; retreatment
MeSH Terms: interventions — mirabegron

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women received Mirabegron: Women with overactive bladder syndrome received Mirabegron
  Interventions: Drug: Mirabegron 25mg

INTERVENTIONS:
Drug: Mirabegron 25mg — Mirabegron 25 mg per day
  Other Names: Betmiga

SUMMARY:
Recurrence of female overactive bladder syndrome (OAB) is not uncommon. It is important to decrease the recurrence of female OAB. However, factors predicting recurrence of female OAB, especially for those women who need retreatment is undetermined. Thus, the aim of this study was to elucidate factors predicting retreatment of female OAB.

DETAILED DESCRIPTION:
The medical records, including pad testing, urodynamic studies, lower urinary tract symptoms related questionnaires and bladder diaries of all consecutive women with OAB, who visited urogynecologic clinics in a tertiary referral center, were reviewed. Persistence interval was defined from the date of prescription of mirabegron to the date of discontinuation of mirabegron treatment. Statistical analysis was performed with Kaplan-Meier estimator. Multivariable Cox proportional-hazard model with all variables with p < 0.25 in the univariate analysis was performed to predict OAB retreatment probability.

ELIGIBILITY:
Inclusion Criteria:

* Women with overactive bladder syndrome
* Women complete urodynamic study and bladder diary

Exclusion Criteria:

* Pregnant women
* Incomplete data
* Loss of follow-up
* Acute or chronic urinary tract infection

Ages: 20 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with overactive bladder syndrome who completed urodynamic study and bladder diary and received Mirabegron 25 mg per day
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Recurrent OAB | January 2015 to July 2019
  Recurrent OAB with needs to retreatment

CONTACTS AND LOCATIONS:
Overall Officials: Ho-Hsiung Lin, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
IPD will be shared under reasonable request

REFERENCES:
- [Result] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN; International Urogynecological Association; International Continence Society. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Neurourol Urodyn. 2010;29(1):4-20. doi: 10.1002/nau.20798. PMID 19941278
- [Result] Coyne KS, Wein AJ, Tubaro A, Sexton CC, Thompson CL, Kopp ZS, Aiyer LP. The burden of lower urinary tract symptoms: evaluating the effect of LUTS on health-related quality of life, anxiety and depression: EpiLUTS. BJU Int. 2009 Apr;103 Suppl 3:4-11. doi: 10.1111/j.1464-410X.2009.08371.x. PMID 19302497
- [Result] Hsiao SM, Lin HH. Medical treatment of female overactive bladder syndrome and treatment-related effects. J Formos Med Assoc. 2018 Oct;117(10):871-878. doi: 10.1016/j.jfma.2018.01.011. Epub 2018 Feb 15. PMID 29398096
- [Result] Hsiao SM, Su TC, Chen CH, Chang TC, Lin HH. Autonomic dysfunction and arterial stiffness in female overactive bladder patients and antimuscarinics related effects. Maturitas. 2014 Sep;79(1):65-9. doi: 10.1016/j.maturitas.2014.06.001. Epub 2014 Jun 20. PMID 25022469
- [Result] Hsiao SM, Liao SC, Chen CH, Chang TC, Lin HH. Psychometric assessment of female overactive bladder syndrome and antimuscarinics-related effects. Maturitas. 2014 Dec;79(4):428-34. doi: 10.1016/j.maturitas.2014.08.009. Epub 2014 Sep 3. PMID 25238744
- [Result] Hsiao SM, Chang TC, Chen CH, Wu WY, Lin HH. Frequent nocturia episodes, a suboptimal response to treatment, and small bladder capacity predict the need for persistent antimuscarinic therapy or re-treatment after discontinuation of antimuscarinics in female overactive bladder. Menopause. 2017 Jan;24(1):100-104. doi: 10.1097/GME.0000000000000730. PMID 27648660